CLINICAL TRIAL: NCT01442792
Title: Prospective, Multi-center, Randomized, Heparin-controlled Dose-finding Trial to Evaluate the Efficacy and Safety of Rivaroxaban, a Direct Factor Xa Inhibitor, on the Background of Standard Dual Antiplatelet Therapy to Support Elective Percutaneous Coronary Intervention
Brief Title: Exploring the Efficacy and Safety of Rivaroxaban to Support Elective Percutaneous Coronary Intervention
Acronym: X-PLORER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15572; 2011-001094-58 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-09-29 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Disease; Coronary Artery Disease
Keywords: Angioplasty, Balloon, Coronary
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator)
  Interventions: Drug: UFH
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 4 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939) and UFH

INTERVENTIONS:
Drug: UFH — Unfractionated Heparin: 70-100 IU/Kg bolus and adjusted upon activated coagulation time (ACT) 250 300 seconds
  Arms: Arm 1
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 10 mg single dose Rivaroxaban (per os)
  Arms: Arm 2
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 20 mg single dose Rivaroxaban (per os)
  Arms: Arm 3
Drug: Rivaroxaban (Xarelto, BAY59-7939) and UFH — 10 mg single dose Rivaroxaban (per os) followed by bolus 50 IU/Kg unfractionated heparin (UFH)
  Arms: Arm 4

SUMMARY:
Balloon angioplasty (Percutaneous Coronary Intervention (PCI)) is commonly used to treat patients with obstructive coronary artery disease (CAD). Although PCI is highly effective for the management of CAD, it can potentiate an existing prothrombotic state around lesion areas. A certain level of anticoagulation is required to perform planned PCI safely and to minimize the periprocedural risk of thrombosis and its attendant complications, including myocardial ischemia and infarction (heart attack). Many different anti-thrombotic regimens have been investigated and are currently in use. The aim of this study is to explore whether Rivaroxaban, as compared to unfractionated heparin, on the background of standard dual antiplatelet therapy, can effectively suppress thrombosis and related adverse ischemic events, upon balloon inflation and stent expansion, during elective PCI, without increasing bleeding. The treatment assignment will be done in a semi-blinded design, eg, no blinding for randomization either to Rivaroxaban (one of the three arms) or the control (UFH) group. However, all will be blinded for the treatment dose of rivaroxaban (either 10mg or 20 mg).The 10 mg rivaroxaban plus 50 IU UFH arm will not be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 years or more with no upper age limit and willing to comply with the protocol
* Symptomatic coronary artery disease due to undergo an elective (non-emergent) Percutaneous Coronary Intervention (PCI) on one or two lesions in the native coronary vessel(s). Cardiac standard troponin at baseline is within the normal limits

Exclusion Criteria:

* Conditions that may increase the risk of the PCI procedure
* Conditions that may increase the risk of bleeding
* Significant valvular heart disease
* Calculated creatinine clearance ≤30 mL/min
* Current use of anticoagulant drugs including Vitamin K antagonist (VKA), factor IIa or factor XA inhibitors
* Chronic treatment with non-steroidal anti-inflammatory drugs (NSAIDs)
* Chronic treatment with aspirin > 100mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2013-01-29 (Actual); Study Completion 2013-03-04 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who require bail-out anticoagulant therapy in the context of an ischemic coronary event | During the index Percutaneous Coronary Intervention procedure
The percentage of subjects who experience an angiographic flow limiting thrombotic event | During the index Percutaneous Coronary Intervention procedure
The percentage of subjects who experience thrombus formation on the Percutaneous Coronary Intervention equipment | During the index Percutaneous Coronary Intervention procedure
The percentage of subjects who experience an Myocardial Infarction due to the Percutaneous Coronary Intervention equipment procedure | During the index Percutaneous Coronary Intervention procedure

SECONDARY OUTCOMES:
Bleeding (Thrombolysis in Myocardial Infarction major, minor and Bleeding academic research consortium type 2, 3 and 5) | Up to 30 days post index Percutaneous coronary intervention procedure
Composite of clinical ischemic events (all death, non-fatal Myocardial Infarction, non-fatal stroke and target lesion revascularization | Up to 30 days post index Percutaneous coronary intervention procedure
Coagulation profile of Rivaroxaban (Activated Partial Thromboplastin Time) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Coagulation profile of Rivaroxaban (Prothrombin time) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Coagulation profile of Rivaroxaban (Thrombin Time) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Coagulation profile of Rivaroxaban (Prothrombin Fragment 1+2) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Coagulation profile of Rivaroxaban (Thrombin Anti-thrombin III Complexes) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Coagulation profile of Rivaroxaban (Anti-Xa Activity) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Coagulation profile of Rivaroxaban (endogenous thrombin potential) | 1 to 5 days prior percutaneous coronary intervention (PCI) and the day of PCI (from 2-4 h pre PCI until 48h post PCI or discharge of patient if earlier)
Plasma concentration of Rivaroxaban | The day of percutaneous coronary intervention (PCI) (from 2 to 4 hours before to 6-8 hours after PCI)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Belgium (3):
  - Hasselt
  - Liège
  - Roeselare
- Netherlands (3):
  - Amsterdam
  - Eindhoven
  - Zwolle

REFERENCES:
- [Result] Vranckx P, Leebeek FW, Tijssen JG, Koolen J, Stammen F, Herman JP, de Winter RJ, van T Hof AW, Backx B, Lindeboom W, Kim SY, Kirsch B, van Eickels M, Misselwitz F, Verheugt FW. Peri-procedural use of rivaroxaban in elective percutaneous coronary intervention to treat stable coronary artery disease. The X-PLORER trial. Thromb Haemost. 2015 Aug;114(2):258-67. doi: 10.1160/TH15-01-0061. Epub 2015 Apr 30. PMID 25925992
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/